CLINICAL TRIAL: NCT02831920
Title: CEUS Targeted Biopsies Compared to mpMRI Targeted and Systematic Biopsies for the Detection of Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. ir. H. Wijkstra, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METC 2015_263
Record Dates: First submitted 2016-07-05; First posted 2016-07-13 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
Keywords: Prostate Cancer; MRI; CEUS; Contrast Ultrasound; Fusion; targeted biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): every patient undergoes mpMRI and targeted biopsies, CEUS and targeted biopsies and systematic biopsies. Every patient is therefore its own control.
  Interventions: Other: CEUS and targeted biopsies; Other: MRI and targeted biopsies

INTERVENTIONS:
Other: CEUS and targeted biopsies
Other: MRI and targeted biopsies

SUMMARY:
The current standard for Prostate Cancer (PCa) detection remains taking 10-12 systematic biopsies of the prostate. This approach leads to overdiagnosis of insignificant PCa on the one hand and underdiagnosis and undergrading of significant PCa on the other. multiparametric Magnetic Resonance Imaging (mpMRI) has seen an increasing uptake in the clinics for biopsy targeting, but the value in biopsy naive patients remains controversial. With Contrast Enhanced UltraSound (CEUS) cancer induced neovascularisation can be visualised with the potential to improve ultrasound imaging for prostate cancer detection and localisation significantly. The past years numerous studies have been performed with CEUS, all basing their results on subjective judgement of the investigator. To overcome these difficulties CEUS quantification techniques have been used with encouraging first results. These imaging techniques have been proposed to improve the yield of prostate biopsies and possibly replacing systematic biopsies.

In this trial mpMRI imaging and CEUS + quantification are performed before primary biopsy. Using a fusion device, targeted biopsies are taken from predefined MRI lesions and CEUS lesions, together with standard systematic biopsies in the same patients by separate blinded clinicians. The main outcome measure is the per-patient (significant) prostate cancer detection rate for each of the biopsy regimens.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* signed informed consent
* referred for mpMRI and primary biopsy

Exclusion Criteria:

* Documented acute prostatitis or urinary tract infections
* History of any clinically evidence of cardiac right-to-left shunts
* Receives treatment that includes dobutamine
* Severe pulmonary hypertension (pulmonary artery pressure >90 mmHg) or uncontrolled systemic hypertension or respiratory distress syndrome
* Has received a biopsy procedure within 30 days before admission into this study
* Has received a biopsy procedure at the Academic Medical Center within a year before admission into this study
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study
* Is incapable of understanding the language in which the information for the patient is given

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Estimated)
Dates: Start 2015-12-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
per-patient (significant) prostate cancer detection rate of mpMRI targeted biopsies | 2 weeks
per-patient (significant) prostate cancer detection rate of CEUS targeted biopsies | 2 weeks
per-patient (significant) prostate cancer detection rate of systematic biopsies | 2 weeks

SECONDARY OUTCOMES:
complementarity of CEUS and mpMRI targeted biopsies in terms of per-patient (significant) cancer detection rate | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hessel H. Wijkstra, Prof dr ir, Principal Investigator — AMC University Hospital
Locations (1):
- AMC University Hospital, Amsterdam, Netherlands

REFERENCES:
- [Derived] Butler MB, Papageorgiou G, Kanoulas ED, Voulgaridou V, Wijkstra H, Mischi M, Mannaerts CK, McDougall S, Duncan WC, Lu W, Sboros V. Mapping of prostate cancer microvascular patterns using super-resolution ultrasound imaging. Eur Radiol Exp. 2025 Feb 20;9(1):25. doi: 10.1186/s41747-025-00561-6. PMID 39976631
- [Derived] Postema AW, Scheltema MJ, Mannaerts CK, Van Sloun RJ, Idzenga T, Mischi M, Engelbrecht MR, De la Rosette JJ, Wijkstra H. The prostate cancer detection rates of CEUS-targeted versus MRI-targeted versus systematic TRUS-guided biopsies in biopsy-naive men: a prospective, comparative clinical trial using the same patients. BMC Urol. 2017 Apr 5;17(1):27. doi: 10.1186/s12894-017-0213-7. PMID 28381220